CLINICAL TRIAL: NCT04792476
Title: High Intensity Interval Training to Prevent Weight Gain in Patients With a First-episode Psychosis: a Randomized Clinical Trial
Brief Title: HIIT in Patients With a First-episode Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Intervención Temprana en Psicosis de Cantabria (ITPCan) (Other)
Responsible Party: Principal Investigator, Jose Antonio Cortés Fernández, Principal Investigator, Intervención Temprana en Psicosis de Cantabria (ITPCan)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ITPCan
Record Dates: First submitted 2021-02-28; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: First-episode Psychosis
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Experimental group (Active Comparator): The experimental group will receive, in addition to the conventional treatment, a physical exercise intervention along 12 weeks, which will consist of complying with the general recommendations for physical activity: 75 minutes weekly of high intensity physical exercise. The therapeutic exercise intervention will be supervised by a physiotherapist and designed in a progressive, structured and personalized way.
  Interventions: Other: High Intensity Interval Training
- No Intervention: Control group (No Intervention): The control group will only receive the conventional treatment offered in the clinical program. For 12 weeks, parients will attend 8 visits with mental health specialist nurse, where they will receive information, oral and written, to comply with the recommendations for physical exercise: 150-300 min/week of moderate physical activity or 75-150 min/week of vigorous physical activity.
  In both groups (experimental and control), patients will be informed of the risk of weight gain, and they will be advised, regardless of the group assigned, to watch their diet and increase physical exercise until they meet the weekly recommendations.

INTERVENTIONS:
Other: High Intensity Interval Training — Experimental group will receive, in addition to the conventional treatment, a physical exercise intervention along 12 weeks, which will consist of complying with the general recommendations for physical activity: 75 minutes weekly of high intensity physical exercise. The therapeutic exercise intervention will be supervised by a physiotherapist and designed in a progressive, structured and personalized way.
  Arms: Active Comparator: Experimental group

SUMMARY:
This study aims to estimate the effect of a 3-month High Intensity Interval Training on antipsychotic-induced weight gain in patients with a first episode of psychosis, as well as to determine whether these effects are maintained 9 months after the intervention has ended.

DETAILED DESCRIPTION:
Weight gain associated with antipsychotic medication has been recognized for years as a very common side effect, occurring mainly during the first months after the start of antipsychotic treatment. Patients with schizophrenia have a risk of obesity 1.5-2 times higher than the general population and the chances of developing physical problems such as hypertension, diabetes, metabolic syndrome, and coronary heart disease are also higher. Patients diagnosed with schizophrenia have a life expectancy of up to 25 years lower than the general population, with cardiovascular disease being the main cause of premature death. The first months of treatment constitute a critical period for the implementation of strategies that could prevent or mitigate this side effect of the medication, as well as the adverse consequences derived from weight gain.

This project is the response to the need to implement physical exercise interventions to prevent weight gain in patients with a first psychotic episode.To date, there is little evidence from randomized clinical trials that have used physical exercise as the only intervention to prevent weight gain in the first weeks from the start of antipsychotic treatment.

Numerous systematic reviews and meta-analyses have evaluated non-pharmacological interventions to reduce weight in people with severe mental illness, including chronic psychotic disorders. However, there is little research on this type of intervention in patients with a first episode of psychosis. Studies are needed that implement physical exercise programs from the initial phases of antipsychotic treatment, and that are capable of defining the parameters used in the design of an effective physical exercise intervention for the prevention of weight gain in first psychotic episodes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤40 years.
* Treatment with antipsychotic medication ≤6 weeks.
* Diagnosis of First Episode Psychosis, for inclusion in the ITPCan Clinical Program.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Poorly controlled diabetes.
* Moderate or severe intellectual disability.
* Current High Intensity Interval Training program.
* Any systematic disease that contraindicates High Intensity Interval Training.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight gain induced by antipsychotic treatment in patients with a first episode of psychosis with a 12-week High Intensity Interval Training. | 12 weeks
Change in weight gain induced by antipsychotic treatment in patients with a first episode of psychosis at 9 months after finishing the intervention. | 9 months post-intervention

SECONDARY OUTCOMES:
Change in the lipid metabolism: triglycerides levels, total cholesterol levels, HDL cholesterol levels and LDL cholesterol levels. | 12 weeks and 9 months post-intervention
  Dyslipidemia is an abnormal amount of lipids (e.g.,triglycerides, cholesterol and/or fat phospholipids) in the blood.
  The normal triglyceride level is between 30 and 150 mg/dL. The normal HDL cholesterol level is between 40 and 60 mg/dL.
Change in abdominal obesity measured by waist circumference. | 12 weeks and 9 months post-intervention
  Abdominal obesity, also known as central obesity, is when excessive abdominal fat around the stomach and abdomen has built up to the extent that it is likely to have a negative impact on health.
  Men are considered to be at high risk from abdominal obesity if their waist measurements are 102 cm or higher, while women are considered to be at high risk if their waist measurements are 88 cm or higher.
Change in glycemic measured by fasting plasma glucose, glycosylated hemoglobin HbA1c and insulin. | 12 weeks and 9 months post-intervention
  Hyperglycemia, or high blood sugar (also spelled hyperglycaemia) is a condition in which an excessive amount of glucose circulates in the blood plasma.
  A subject with a consistent range between 100-126 mg/dl is considered hyperglycemic, while above 126 mg/dl is generally held to have diabetes.
Change in hypertension measured by blood pressure. | 12 weeks and 9 months post-intervention
  Hypertension (HTN or HT), also known as high blood pressure (HBP), is a long term medical condition in which the blood pressure in the arteries is persistently elevated.
  Blood pressure is expressed by two measurements, the systolic and diastolic pressures, which are the maximum and minimum pressures, respectively. Normal blood pressure at rest is within the range of 100-130 millimeters mercury (mmHg) systolic and 60-85 mmHg diastolic.

IPD SHARING:
Plan to Share IPD: No